CLINICAL TRIAL: NCT06816043
Title: An Open-label, Phase 1 Study to Characterize the Effects of Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) on the Pharmacokinetics of MK-8527 in Healthy Participants
Brief Title: A Study of Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) and MK-8527 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 8527-016; MK-8527-016 (Other: MSD)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: MK-8527 (Experimental): Participants receive a single dose of MK-8527.
  Interventions: Drug: MK-8527
- Treatment B: MK-8527 + FTC/TDF (Experimental): Participants receive FTC/TDF then MK-8527.
  Interventions: Drug: MK-8527; Drug: FTC/TDF

INTERVENTIONS:
Drug: MK-8527 — Oral Capsule
Drug: FTC/TDF — Oral Tablet
  Other Names: emtricitabine/tenofovir disoproxil fumarate
  Arms: Treatment B: MK-8527 + FTC/TDF

SUMMARY:
The goal of this study is to learn what happens to MK-8527 in a healthy person's body over time, called a pharmacokinetic (PK) study. Researchers want to learn if there is a difference in the healthy person's body when MK-8527 is taken as a single dose (Treatment A) or with the medication Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) (Treatment B).

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior
* Has body mass index (BMI) ≥18 and ≤32.0 kg/m^2

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History of low bone density, renal impairment, Fanconi syndrome, autoimmune disorders (such as Graves' disease, polymyositis, Guillain-Barré syndrome, and autoimmune hepatitis), liver disease
* History of cancer (malignancy)
* Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity after single dosing (AUC0-Inf) of MK-8527-Triphosphate (TP) in peripheral blood mononuclear cell (PBMC) | Pre-dose and at designated time points up to 840 hours post dose
  Blood samples will be collected to determine the AUC0-Inf of MK-8527-TP in PBMC.
Area Under the Concentration-Time Curve from Time 0 to Last quantifiable sample (AUC0-last) of MK-8527-TP in PBMC | Pre-dose and at designated time points up to 840 hours post dose
  Blood samples will be collected to determine the AUC0-last of MK-8527-TP in PBMC.
Drug Concentration at 672 Hours (C672) of MK-8527-TP in PBMC | Pre-dose and at designated time points up to 672 hours post dose
  Blood samples will be collected to determine the C672 of MK-8527-TP in PBMC.
Maximum Plasma Concentration (Cmax) of MK-8527-TP in PBMC | Pre-dose and at designated time points up to 840 hours post dose
  Blood samples will be collected to determine the Cmax of MK-8527-TP in PBMC.
Time to Maximum Plasma Concentration (Tmax) of MK-8527-TP in PBMC | Pre-dose and at designated time points up to 840 hours post dose
  Blood samples will be collected to determine the Tmax of MK-8527-TP in PBMC.
Apparent Terminal Half-life (t1/2) of MK-8527-TP in PBMC | Pre-dose and at designated time points up to 840 hours post dose
  Blood samples will be collected to determine the t1/2 of MK-8527-TP in PBMC.

SECONDARY OUTCOMES:
AUC0-Inf of MK-8527 in plasma | Pre-dose and at designated time points up to 120 hours post dose
  Blood samples will be collected to determine the AUC0-Inf of MK-8527 in plasma.
AUC0-last of MK-8527 in plasma | Pre-dose and at designated time points up to 120 hours post dose
  Blood samples will be collected to determine the AUC0-last of MK-8527 in plasma.
Cmax of of MK-8527 in plasma | Pre-dose and at designated time points up to 120 hours post dose
  Blood samples will be collected to determine the Cmax of MK-8527 in plasma.
Tmax of MK-8527 in plasma | Pre-dose and at designated time points up to 120 hours post dose
  Blood samples will be collected to determine the Tmax of MK-8527 in plasma.
t1/2 of MK-8527 in plasma | Pre-dose and at designated time points up to 120 hours post dose
  Blood samples will be collected to determine the t1/2 of MK-8527 in plasma.
Apparent Clearance (CL/F) of MK-8527 in plasma | Pre-dose and at designated time points up to 120 hours post dose
  Blood samples will be collected to determine the CL/F MK-8527 in plasma
Apparent volume of distribution during terminal phase (Vz/F) of MK-8527 in plasma | Pre-dose and at designated time points up to 120 hours post dose
  Blood samples will be collected to determine the Vz/F of MK-8527 in plasma
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 111 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 43 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com